CLINICAL TRIAL: NCT05923671
Title: Clinical, Histological and Immunohistochemical Characterization of Human Gingival Phenotypes
Brief Title: Clinical and Histological Analysis of Human Gingival Phenotypes
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 1399
Record Dates: First submitted 2023-03-22; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: gingiva; histological; immunohistochemical; periodontal; biotype; phenotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thin Phenotype: Participants with transparent free gingiva of the maxillary central incisor
  Interventions: Diagnostic Test: Histological analysis; Diagnostic Test: Immunohistochemical analysis
- Thick Phenotype: Participants with non-transparent free gingiva of the maxillary central incisor
  Interventions: Diagnostic Test: Histological analysis; Diagnostic Test: Immunohistochemical analysis

INTERVENTIONS:
Diagnostic Test: Histological analysis — Histological staining of gingival biopsies with haematoxylin-eosin.
Diagnostic Test: Immunohistochemical analysis — Immunohistochemical staining of gingival biopsies using anti-Vimentin, anti-Collagen I, anti-Collagen V, anti-Elastin, anti-Hyaluronic acid, anti-Smooth muscle actin, anti-Cluster of Differentiation 68 and anti-ki67 antibodies.

SUMMARY:
The goal of this observational study is to compare the composition of the human gingiva in different gingival phenotypes. The main questions to answer are:

* Is there any difference in the cellular composition of the gingiva between thin and thick gingival phenotype?
* Is there any difference in the molecular composition of the gingiva between thin and thick gingival phenotype?

The participants were divided in two groups (thin and thick phenotype) and a biopsy of healthy gingiva was obtained from each one them. The biopsies were analyzed histologically and the collected data will be analyzed statistically in order to identify possible differences between the gingival phenotypes.

DETAILED DESCRIPTION:
Healthy volunteers were assigned in one of two groups:

* Group 1: Thin gingiva, when the free gingiva was evaluated as transparent, after the insertion of a periodontal probe (Hu-Friedy XP-23/QW, Hu-Friedy,Chicago,IL,USA) in the middle of the facial dentogingival sulcus of a maxillary central incisor
* Group 2: Thick gingiva: when the free gingiva was evaluated as non-transparent, using the same methodology.

A full thickness sample of the oral mucosa of each one of the participants was collected under local anaesthesia. The sample had a rectangular shape, with a length of 4 millimeters and a width of 1 millimeter. It had a vertical orientation and it was expanding at the both sides of the mucogingival junction.

The oral mucosa samples were processed for histological and immunohistochemical analysis. Staining with haematoxylin-eosin was performed in order to describe the tissue histologically and also calculate the total number of the cells it contained. Immunohistochemical staining with anti-Vimentin,anti-Cluster of Differentiation 68, anti-Ki-67 and anti-Smooth Muscle Actin antibodies was applied for the calculation of the numbers of fibroblasts, macrophages, Ki-67-positive cells and Smooth muscle actin positive cells respectively. Immunohistochemical staining was also performed in order to determine the levels of expression of Collagen I, Collagen V, Elastin and Hyaluronic acid.

Whole slide images of the specimens were acquired with the use of the NanoZoomer 2.0HT (Hamamatsu Pho-tonics K.K., Hamamatsu, Japan). Cell counting will be performed automatically using an image analysis software (QuPath 3.0). The levels of molecular expression will be assessed with the use of the same software and will be expressed as a percentage of the area of the connective tissue that is occupied by the investigated molecules.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Attachment loss or Probing depths greater than 2 millimeters at the maxillary central incisors
* Altered passive eruption of the maxillary incisors
* Previous surgery or orthodontic treatment in the anterior maxilla
* Medical conditions or medication affecting soft tissue metabolism
* Tooth crowding or abnormal angulation or abrasion of the maxillary incisors
* Restorations at the buccal surface of the maxillary central incisors
* Smoking
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers referred to the Department of Preventive Dentistry, Periodontology and Implant Biology of the Dental School of the Aristotle University of Thessaloniki.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Cell density | Baseline
  The number of all types of cells per square millimeter of the connective tissue

SECONDARY OUTCOMES:
Fibroblast Density | Baseline
  The number of fibroblasts per square millimeter of the connective tissue
Macrophage Density | Baseline
  The number of macrophages per square millimeter of the connective tissue
Density of Ki-67-positive cells | Baseline
  The number of Ki-67-positive cells per square millimeter of the connective tissue
Density of Smooth Muscle Actin positive cells | Baseline
  The number of Smooth Muscle Actin positive cells per square millimeter of the connective tissue
Collagen I area ratio | Baseline
  The percentage of the area of the connective tissue which is occupied by Collagen I
Collagen V area ratio | Baseline
  The percentage of the area of the connective tissue which is occupied by Collagen V
Elastin area ratio | Baseline
  The percentage of the area of the connective tissue which is occupied by Elastin
Hyaluronic acid area ratio | Baseline
  The percentage of the area of the connective tissue which is occupied by Hyaluronic acid

OTHER OUTCOMES:
Keratinized tissue width | Baseline
  The length (millimeters) of the line that connects the mucogingival junction and the gingival margin, at the middle of the facial surface of the maxillary central incisor
Gingival thickness | Baseline
  The thickness (millimeters) of the gingiva, measured with an ultrasonic biometer (PIROP Biometric scanner, ECHO-SON S.A., Poland) at the middle of the line that connects the mucogingival junction and the gingival margin, at the middle of the facial surface of the maxillary central incisor

CONTACTS AND LOCATIONS:
Overall Officials: Sotiris Kalfas, Professor, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Macedonia, Greece